CLINICAL TRIAL: NCT04832815
Title: Equine Human Interaction With Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Collaborators: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00125426
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: PTSD
Keywords: Equine; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Equine Therapy (Experimental)
  Interventions: Behavioral: Equine Therapy
- Treatment as Usual (TAU) (No Intervention)
- Therapeutic Horsemanship Program (Experimental)
  Interventions: Behavioral: Therapeutic Horsemanship Program

INTERVENTIONS:
Behavioral: Equine Therapy — Aim 1: Six session equine interventions. Intervention will be provided one day per week for four weeks. During the first two weeks, each intervention day with consist of two sessions with a lunch break in between. Weeks four and five consist of one trail riding session per intervention day followed by lunch. Each session will be approximately 1.5 hours in length. Sessions 1-4 will occur at the USU Equine Education Center, and session 5-6 will occur on local trails. Optional transportation for participants will be provided from the VA to the intervention site.
  Arms: Equine Therapy
Behavioral: Therapeutic Horsemanship Program — Aim 2: Therapeutic Horsemanship program utilizes the USU Pathways to Horsemanship model and covers levels of equestrian training from basic groundwork to more advanced riding techniques. Training occurs in a three or six-session format with once weekly sessions over three or six weeks. Mindfulness and mindful self-compassion training may be included.
  Arms: Therapeutic Horsemanship Program

SUMMARY:
This study has two components. The first component (Aim 1) is a randomized trial of a novel equine therapy intervention that was developed for research purposes. The second component (Aim 2) is an evaluation of outcomes from Veterans participating in an adaptive horsemanship program that is not conducted for research purposes.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1:

* Currently enrolled for services at the VA Salt Lake City Health Care System
* At least one mental health service encounter within the preceding 12 months
* Diagnosed with PTSD by a clinician within the preceding 24 months
* Have a doctor release to participate in equine activities

For Aim 2:

* Currently enrolled for services at the VA Salt Lake City Health Care System
* Have a doctor release to participate in equine activities

Exclusion Criteria:

* Pregnancy
* Diagnoses of a psychotic spectrum illness and/or cognitive impairment
* Physical disability that would prevent horseback riding
* Weight >= 250 lbs.
* Potentially the severity of and psychological and/or behavioral symptoms will be considered

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-12-19 (Estimated); Study Completion 2024-12-19 (Estimated)

PRIMARY OUTCOMES:
Mean Difference in Acceptance and Action Questionnaire-II (AAQII) among the Equine Therapy + TAU cohort compared to the TAU only cohort and for Horsemanship Skills Training Program | through study completion, an average of 2 years
  AAQII measures psychological flexibility. The total AAQII score can range from 7 to 49, with higher values indicating greater psychological inflexibility. Mixed Effect Modeling will be used for the analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate the outcome at multiple time points: pre-intervention, post-intervention for selected or all sessions, and post-intervention.
Heart Rate (HR) Indices | through study completion, an average of 2 years
  To determine correlations between physiological responses of the rider and horse, the following heart rate (HR) indices will be computed: Mean HR, standard deviation of the beat-to-beat intervals (SDRR) and the root mean square of successive beat-to-beat differences (rMSSD). Both SDRR and rMSSD are measures of HR variability and reflect shifts between sympathetic (e.g., decrease in HR variability) or parasympathetic (e.g., increase in HR variability) drive. These measures will be taken during each equine intervention session.
Mean Difference in Positive and Negative Affect Scale (PANAS) among the Equine Therapy + TAU cohort compared to the TAU only cohort and for Horsemanship Skills Training Program | through study completion, an average of 2 years
  PANAS measures short-term positive and negative emotions. The total PANAS-C score can range from 12 to 60 for the positive affect (PA) scale, with higher values indicating greater PA. Similarly, the score range from 15 to 75 for the negative affect (NA) scale, with higher values indicating greater NA. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate the primary outcome at multiple time points: pre-intervention, post-intervention sessions, and post-intervention.
Mean Difference in Physical Activity Enjoyment Scale (PACES) for Equine Therapy + TAU cohort compared to the TAU only cohort and for Horsemanship Skills Training Program | through study completion, an average of 2 years
  PACES measures enjoyment of activity. The total PACES score can range from 18 to 126, with higher values indicating greater enjoyment. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate the outcome after the intervention sessions and post-intervention.
Mean Difference in Posttraumatic Stress Disorder Checklist (PCL) for Equine Therapy + TAU cohort compared to the TAU only cohort | through study completion, an average of 2 years
  PCL measures PTSD symptoms. The total PCL score can range from 17 to 85, with higher values indicating greater PTSD symptoms. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate outcome post-intervention sessions and post-intervention.
Mean Difference in Beck Depression Inventory (BDI) for Equine Therapy + TAU cohort compared to the TAU only cohort | through study completion, an average of 2 years
  BDI measures depressive symptoms. The total BDI score can range from 0 to 63, with higher values indicating greater depressive symptoms. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate outcome post-intervention sessions and post-intervention.
Mean Difference in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) for Horsemanship Skills Training Program and for Equine Therapy + TAU cohort compared to the TAU only cohort | through study completion, an average of 2 years
  Q-LES-Q-SF measures quality of, and satisfaction with, life. The total Q-LES-Q-SF score can range from 14 to 70, with higher values indicating greater satisfaction. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate outcome post-intervention sessions and post-intervention.
Mean and Standard Deviation of Personal Satisfaction Program Survey for Horsemanship Skills Training Program and for Equine Therapy + TAU cohort compared to the TAU only cohort | through study completion, an average of 2 years
  Personal Satisfaction Program Survey measures satisfaction with the program. The total Personal Satisfaction Program Survey score can range from 0 to 210, with higher values indicating greater program satisfaction. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate outcome post-intervention sessions and post-intervention.
Mean Difference in Toronto Mindfulness Scale (TMS) for Equine Therapy + TAU cohort | through study completion, an average of 2 years
  TMS measures state mindfulness. The total TMS score can range from 0 to 52, with higher values indicating greater state mindfulness. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate outcome pre-intervention, post-intervention sessions, post-intervention.
Mean Difference in Five Facet Mindfulness Questionnaire (FFMQ) for Horsemanship Skills Training Program. | through study completion, an average of 2 years
  The total FFMQ score can range from 8 to 40 for each of the facets (observe, describe, act aware, nonjudge, nonreact), with higher values indicating greater levels of mindfulness. Mixed Effect Modeling will be used for the primary analyses. Within and between group analyses of pre- to post-intervention psychological instrument and service utilization data will be conducted to determine whether outcomes are associated with program participation. We'll estimate outcome post-intervention.

SECONDARY OUTCOMES:
Mean and Standard Deviation of Demographic information including medical and psychiatric diagnoses | through study completion, an average of 2 years
  Demographic information as well as medical and psychiatric diagnoses of the participants will be extracted from the electronic medical record. Demographic information includes age, race, ethnicity, and service connection.
  Numbers of psychiatric hospitalizations and emergency department visits for 6 months pre- and 6 months post-intervention will be extracted from the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: William R Marchand, MD, Principal Investigator — Salt Lake City Veterans' Administration Medical Center
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No